CLINICAL TRIAL: NCT03803657
Title: Comparison of Measured Caloric Expenditure Versus Administered Calories in Neonates
Status: Withdrawn | Type: Observational
Why Stopped: Never started
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John Kheir, Staff physician, Boston Children's Hospital
Other Study IDs: IRB-P00030228
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Calorie Overload; Calorie Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Neonates: Neonates 0-28 days
  Interventions: Device: Monitoring of energy expenditure
- Infant: 29 days to 1 year
  Interventions: Device: Monitoring of energy expenditure
- Child: >1 year and <10 kg
  Interventions: Device: Monitoring of energy expenditure

INTERVENTIONS:
Device: Monitoring of energy expenditure — Continuous monitoring of energy expenditure.

SUMMARY:
The investigators have created and validated a device that allows us to accurately measure how many calories a baby consumes every day. The purpose of this study is to compare how many calories a baby consumes with how many calories are provided in a population of newborn infants and children. This may help clinicians to better understand how to feed babies during times of critical illness.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanically ventilated neonates, infants and children, regardless of age, up to 10 kg
2. Inpatients in the cardiac (8S), medical-surgical (7S) or neonatal (7N) intensive care unit
3. Assent of patient's intensive care attending physician
4. Written parental informed consent.
5. Patient on conventional mechanical ventilation on a Servo I or Servo U ventilator with fraction of inspired oxygen <80%.

Exclusion Criteria:

1. Clinically significant tracheo-esophageal fistula
2. Measured ETT leak >20% (i.e. difference between inspiratory and expiratory tidal volumes)
3. Patient on high frequency oscillatory ventilation or high frequency jet ventilation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mechanically ventilated children.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Average caloric expenditure | through study completion, an average of 3 days
  Number of calories consumed

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nachman E, Clemensen P, Santos K, Cole AR, Polizzotti BD, Hofmann G, Leeman KT, van den Bosch SJ, Kheir JN. A Device for the Quantification of Oxygen Consumption and Caloric Expenditure in the Neonatal Range. Anesth Analg. 2018 Jul;127(1):95-104. doi: 10.1213/ANE.0000000000003308. PMID 29505450